CLINICAL TRIAL: NCT01459250
Title: An Open Label, Non-randomised, Parallel Group Study to Characterise and Compare the Pharmacokinetics, Safety and Tolerability of a Single Dose of AGO178C in Subjects With Mild, Moderate, Severe Renal Impairment and End-stage Renal Disease With That in Healthy Matched Control Subjects
Brief Title: Pharmacokinetics, Safety and Tolerability of AGO178C in Subjects With Renal Deficiencies Compared With Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAGO178C2104
Record Dates: First submitted 2011-09-23; First posted 2011-10-25 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2011-10

CONDITIONS: Renal Impairment
Keywords: AGO178C,; renal impairment,; ESRD,; pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic

ARMS (1):
- AGO178C (Experimental)
  Interventions: Drug: AGO178C

INTERVENTIONS:
Drug: AGO178C

SUMMARY:
This study will assess the pharmacokinetics, safety and tolerability of a single dose of AGO178C in subjects with mild, moderate, severe renal impairment and end-stage renal disease with that in healthy matched control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Mild, moderate, severe renally impaired or ESRD patients.
* Healthy male or female subjects to match renally impaired patients in BMI (±15%), age (± 7 years) and gender (in this order). Smoking status (yes or no) will also be used as a final criterion, if deemed feasible by the Investigator.

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless using effective contraception during the study as defined in the protocol.
* Smokers, smoking 10 cigarettes or more per day from screening to study completion
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study
* Co-medication for healthy subjects

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Measure: Composite of AGO178C pharmacokinetics in blood and urine samples. | pre dose, 2 min, 5 min, 10 min, 20 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 12 h, 24 h and 36 h post dose

SECONDARY OUTCOMES:
Measure: Safety and tolerability of AGO178C as assessed by adverse events reports, vital signs, ECGs and safety laboratory tests. | Up to 9 Days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Knoxville, Tennessee

REFERENCES:
- See also: Results for CAGO178C2104 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6944